CLINICAL TRIAL: NCT00474877
Title: The Clinical Effectiveness of Static Resting Splints in Early Rheumatoid Arthritis: a Randomized Controlled Trial
Brief Title: The Clinical Effectiveness of Static Resting Splints in Early Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MREC/01/6/43
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Clinical; Splints; Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Static resting splints

SUMMARY:
This study tested the hypothesis that there would be a difference in the 12 month progression of structural hand impairment and hand function between a group of patients with early RA who received static resting splints and those that did not.

DETAILED DESCRIPTION:
This study is a multi centred RCT recruiting patients across 8 rheumatology occupational therapy departments in the UK. Patients with early RA (<5 years) were recruited. The study followed patients over a 12 month treatment period. Patients were randomised to receive standardised occupational therapy or standardised occupational therapy plus static resting splints over 12 months. The primary outcome measure was dominant hand grip strength and secondary out measures included; dominant hand MCPJ ulnar deviation, the button board from the Arthritis Hand Function Test and the Michigan Hand Outcomes Questionnaire.

Data were analysed using ANCOVA. Baseline outcome values, Ritchie Scores at baseline and the number of intra articular wrist and hand steroid injections were controlled for as covariates.

This study is a multi centred RCT recruiting patients across 8 rheuamtology occupational therapy departments in the UK. Patients with early RA (<5 years) were recruited. The study followed patients over a 12 month treamtent period. Patients were randomised to receive standardised occupational therapy or standardised occupational therapy plus static resting splints over 12 months. The primary outcome measure was dominant hand grip strength and secondary out measures included; dominant hand MCPJ ulnar deviation, the button board from the Arthritis Hand Function Test and the Michigan Hand Outcomes Questionnaire.

Data were analysed using ANCOVA. Baseline outcome values, Ritchie Scores at baseline and the number of intra articular wirst and hand steroid injections were controlled for as covariates.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of RA, less than 5 years duration

Exclusion Criteria:

* Patients with previous wrist and hand surgery, non-addressable fixed hand or wrist deformity, those from vulnerable group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-10; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Dominant power hand grip (Newtons) | 12 months

SECONDARY OUTCOMES:
MCPJ ulnar deviation | 12 months
Michigan Hand Outcome Questionnaire | 12 months
Applied dexterity - Button Board Arthritis Hand Function Test | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jo E Adams, PhD, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hants, United Kingdom